CLINICAL TRIAL: NCT06635525
Title: IMPACT OF KIDNEY FAILURE ON THE REGULATION OF HUMORAL RESPONSE TO VACCINATION
Acronym: Tfh-CKD
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: Fondazione Cariplo (Unknown)
Responsible Party: Sponsor
Other Study IDs: 5281
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis; Vaccine Response
Keywords: Vaccine; Influenza; Chronic Kidney Disease; Hemodialysis; Peritoneal dialysis; Humoral Response
MeSH Terms: conditions — Influenza, Human; Renal Insufficiency, Chronic | interventions — Influenza Vaccines; COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hemodialysis patients: Subjects with advanced chronic kidney disease requiring thrice-weekly hemodialysis
  Interventions: Biological: Influenza vaccination; Biological: SARS-CoV-2 vaccine
- Peritoneal dialysis patients: Subjects with advanced chronic kidney disease on peritoneal dialysis
  Interventions: Biological: Influenza vaccination; Biological: SARS-CoV-2 vaccine
- Healthy controls: Subjects without a prior history of chronic kidney disease
  Interventions: Biological: Influenza vaccination; Biological: SARS-CoV-2 vaccine

INTERVENTIONS:
Biological: Influenza vaccination — Single-dose
Biological: SARS-CoV-2 vaccine — Single-dose

SUMMARY:
The aim of this observational study is to determine if and how kidney failure affects the development of protective immune responses following vaccination in patients on chronic dialysis.

Researchers will compare the effectiveness of the influenza vaccine in inducing protective antibodies between hemodialysis patients and subjects without chronic kidney disease.

Participants will:

* Be enrolled at the time of influenza vaccination
* Visit the clinic at 7, 14, 30, 60, and 120 days after vaccination
* Be asked to provide relevant clinical information and a blood sample at each visit

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Patients undergoing thrice-weekly hemodialysis / peritoneal dialysis for at least 3 months OR healthy individuals without a history of renal insufficiency
* Subjects eligible to receive a seasonal influenza vaccine
* Signed informed consent for participation in the study

Exclusion Criteria:

* Recent influenza infection (clinically resolved less than 3 months ago).
* Administration of immunosuppressive drugs in the two weeks prior to vaccination.
* Administration of another vaccine in the three weeks prior to enrollment (co-administration of other vaccines with those under study does not contraindicate participation).
* Systemic infection clinically resolved less than two weeks before enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study populations consist of (1) subjects with advanced chronic kidney disease requiring thrice-weekly hemodialysis, (2) subjects with advanced chronic kidney disease on peritoneal dialysis, and (3) subjects without a prior medical history of chronic kidney disease, who are eligible to receive an influenza vaccine according to standard clinical practice guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Frequency of serological response to influenza vaccination | From enrollment to 30±3 days after vaccination

SECONDARY OUTCOMES:
Titer of influenza-specific antibodies after vaccination | From enrollment to 30±3 days after vaccination
Correlation between virus-specific antibody concentration after influenza vaccination and the frequency of circulating T follicular helper cell subsets | From enrollment to 120±5 days after vaccination
Degree of antigen-specific activation of T follicular helper and B cells in vitro after influenza vaccination | From enrollment to 120±5 days after vaccination
Degree of polyclonal activation of T follicular helper and B cells in vitro after exposure to the serum of subjects vaccinated against influenza | From enrollment to 120±5 days after vaccination
Single-cell transcriptome expression in circulating T follicular helper cell subsets | From enrollment to 120±5 days after vaccination

OTHER OUTCOMES:
SARS-CoV-2-specific antibody concentration after vaccination | From enrollment to 30±3 days after vaccination
Correlation between virus-specific antibody concentration after SARS-CoV-2 vaccination and the frequency of circulating T follicular helper cell subsets | From enrollment to 120±5 days after vaccination
Degree of antigen-specific activation of T follicular helper and B cells in vitro after SARS-CoV-2 vaccination | From enrollment to 120±5 days after vaccination

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - ASST Santi Paolo e Carlo, Milan
  - ASST Fatebenefratelli Sacco, Milan

IPD SHARING:
Plan to Share IPD: Undecided